Study Protocol 09/23/2017

PROTOCOL: MATERIAL AND METHODS Study group: 12 healthy subjects of both sexes, selected according to a sample of criteria, aged between 65 and 85 years, with no diagnosed alterations in the balance Place of assessment: domicile of each subject. Ethical aspects: The application of BESTest in the subject group does not involve any invasive activity. According to the Helsinki Declaration, participants will receive oral and written information from the study and will sign an informed consent model attached. Inclusion criteria: No health problems relating to disturbances of balance. Personal autonomy. Cognitive ability to receive three verbal instructions. Ability to sign informed consent. Ability to walk 6 meters without assistance from another person. Ability to perform the test without excessive fatigue. Exclusion criteria. Subjects with diagnosed balance problems. Drop in the three months prior to the study. Need for orthopedic support for walking. Material: Questionnaire. Chronometer. Measuring tape. Rubber foam approximately 60 x 60 centimeters, 10 cm high and medium density. Ramp with inclination of 10 degrees (at least 60 x 60 cm). Steps 15 centimeters high. Two boxes of shoes stacked. A bag of 2.5 kilograms of weight. Chair with armrests. Scotch tape. Method.1: Translation by gualified persons in Spain of BESTest and Mini BESTest. 2: Retro-translation: by qualified persons, other than those who perform the translation. 3: Review Committee: by a group of experts who perform the cultural adaptation of the test. To ensure that the translation is understandable and verify the cultural equivalence of the new version. 4.Application of the tests: BESTest, MiniBEST test, Berg Balance Scale, Fall Effectiveness Scale Test, Up and go test. Simple blind study. The administration of the tests is carried out by one of the researchers, qualified for its administration. The subjects perform the tests in the same session and in their homes with an approximate duration of 1 hour and a half. To each patient is assigned a code. The data obtained with their assignment code are transferred to the second researcher, blinded about the functional characteristics of the participants, who performs the statistical analysis to obtain results.